CLINICAL TRIAL: NCT05069844
Title: Preoperative Gum Chewing for Different Durations to Prevent Sore Throat After Endotracheal Intubation: A Randomized Controlled Trial
Brief Title: Preoperative Gum Chewing for Different Durations to Prevent Sore Throat After Endotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Salah Ahmed Abd Elgalil (Other)
Responsible Party: Sponsor-Investigator, Ahmed Salah Ahmed Abd Elgalil, Lecturer of Anesthesiology and Pain Management, National Cancer Institute, Egypt
Organization: National Cancer Institute, Egypt (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AP2106-50108
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Gum Chewing; Sore Throat; Endotracheal Intubation; Randomized Controlled Trial
MeSH Terms: conditions — Pharyngitis | interventions — Chewing Gum

STUDY DESIGN:
Intervention Model Description: Patients included in the study will be divided into 3 groups; the gum group2 (group G2), the gum group4 (group G4) and the control group (group C) by a computer-generated random number table before surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gum chewing for 2 minutes (Experimental): Patients will chew 1 piece of herbal sugar-free for 2 minutes and then spat it out.
  Interventions: Dietary Supplement: Gum chewing for 2 minutes
- Gum chewing for 4 minutes (Experimental): Patients will chew 1 piece of herbal sugar-free for 4 minutes and then spat it out.
  Interventions: Dietary Supplement: Gum chewing for 4 minutes
- Control group (No Intervention): Patients will be asked to swallow 2 times only.

INTERVENTIONS:
Dietary Supplement: Gum chewing for 2 minutes — In the preoperative waiting area before transfer to the operating room, patients will chew 1 piece of herbal sugar-free for 2 minutes and then spat it out.
  Arms: Gum chewing for 2 minutes
Dietary Supplement: Gum chewing for 4 minutes — In the preoperative waiting area before transfer to the operating room, patients will chew 1 piece of herbal sugar-free for 4 minutes and then spat it out.
  Arms: Gum chewing for 4 minutes

SUMMARY:
This study aims to evaluate the effect preoperative chewing gums for 2 or 4 minutes on postoperative sore throat after general anesthesia using an endotracheal tube.

DETAILED DESCRIPTION:
Pharmacological measures for attenuating postoperative sore throat (POST) include inhalation of beclomethasone or fluticasone propionate; gargling with azulene sulfonate, aspirin, or ketamine: gargling or spraying benzydamine hydrochloride; intravenous (IV) dexamethasone; oral clonidine; topical or systemic lidocaine; and ingestion of strepsils tablets. Each of these approaches has limitations and variable success rates; thus, no approach has become established in routine clinical use. In the past decade, studies have shown that xylitol in chewing gum may inhibit the growth, metabolism, and polysaccharide production of Streptococcus mutans, which accounts for the highest proportion of the natural flora in the oral cavity. Subsequent biofilm formation reduction may lead to some reduction in the number of bacteria. Furthermore, chewing gum can promote salivary gland secretion, resulting in lubrication and cleansing of the oral cavity. which may decrease postoperative sore throat.

Patients included in the study will be divided into 3 groups; the gum group2 (group G2), the gum group4 (group G4) and the control group (group C) by a computer-generated random number table before surgery. In the preoperative waiting area before transfer to the operating room, patients in group G2 will chew 1 piece of herbal sugar-free for 2 minutes and then spat it out, patients in group G4 will chew 1 piece of herbal sugar-free for 4 minutes and then spat it out, group C will be asked to swallow 2 times only. After entering to the OR patients will be routinely monitored with ECG, Pulse oximetry, and blood pressure then induction of anesthesia will be done using Fentanyl 1 to 2 mcg per kg, propofol 1 to 3 mg per kg, and atracurium 0.6 mg per kg. endotracheal tube size 7.5 will be inserted. volume-controlled ventilation was initiated with a mixture of 50% oxygen and 50% air, a respiratory rate of 12 cycles·minute, an inspiratory-to-expiratory ratio (I:E) of 1:2 and an adjusted end-tidal CO2 maintained at approximately 35-40 mm Hg. Ondansetron (4 mg) and paracetamol 1g were injected IV to prevent postoperative nausea, vomiting, and pain. Patients will be extubated after being awake using minimal suction. Postoperative sore throat (POST) will be evaluated by the numerical rating scale (NRS), which ranges from 0 to 10 points, with 0 indicating no pain, 1-3 indicating mild discomfort, 4-6 indicating moderate pain, and 7-10 indicating severe pain.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Age 21-65 years
4. Females
5. American Society of Anesthesiologists (ASA) physical I-II
6. Scheduled for elective breast surgery
7. Under general anesthesia.

Exclusion Criteria:

1. Chronic laryngitis
2. Chronic bronchitis
3. Asthma
4. Gastroesophageal reflux
5. Allergies to study drugs
6. Recent use of nonsteroidal anti-inflammatory drugs (NSAIDs)
7. A history of upper respiratory tract infection
8. Smoking and steroid therapy in the past week
9. Failure to communicate normally
10. Mallampati grade >2

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 150 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
The incidence of moderate/severe postoperative sore throat (POST) within 24 hours after surgery POST within 24 hours after surgery | 24 hours postoperative
  The incidence of moderate/severe POST within 24 hours after surgery

SECONDARY OUTCOMES:
Postoperative sore throat (POST) numeric rating scale (NRS) scores 2, 6, and 24 hours after surgery | 24 hours Postoperative
  POST will be evaluated by the numerical rating scale (NRS), which ranges from 0 to 10 points, with 0 indicating no pain, 1-3 indicating mild discomfort, 4-6 indicating moderate pain, and 7-10 indicating severe pain. The higher is worse.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute - Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP
Time Frame: One year after the end of the study